CLINICAL TRIAL: NCT07052292
Title: DuraTouch® - Post-Market Clinical Follow-up (PMCF) Study in a Real-world Setting
Brief Title: User Experience With DuraTouch® in Patients With Type 1 or Type 2 Diabetes
Status: Active, not recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-8353; U1111-1316-4217 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- DuraTouch® (Insulin injection): Participants will subcutaneously inject the insulin prescribed by the doctor using DuraTouch® according to routine clinical practice at the discretion of the treating physician.
  Interventions: Device: DuraTouch®

INTERVENTIONS:
Device: DuraTouch® — Participants will subcutaneously inject the insulin using DuraTouch®.

SUMMARY:
This study looks at overall impact of the use of DuraTouch® in terms of ease, convenience to use and satisfaction in participants with either type 1 or type 2 diabetes.The study will last for about 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The decision to initiate treatment with DuraTouch® has been made by the participant/legally acceptable representative (LAR) and the treating physician before and independently from the decision to include the participant in this study.
* All needed signed consent(s) are obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Mental incapacity (when no caregiver and LAR are assigned to the patient), unwillingness or language barriers precluding adequate understanding or cooperation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population included participants with Type 1 Diabetes Mellitus (T1DM) or Type 2 Diabetes Mellitus (T2DM) who require insulin injection.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-01-02 (Estimated)

PRIMARY OUTCOMES:
Participant rating the ease of use, convenience and satisfaction with the device | At week 12
  Rating score on a 5-point Likert-type response scale. 1=Not at all easy/convenient/satisfied, 5=Extremely easy/convenient/satisfied.

SECONDARY OUTCOMES:
Participant rating the ease of preparing the device for use and ease of injection | At week 12
  Rating score on a 5-point Likert-type response scale. 1=Not at all easy, 5=Extremely easy.
Participant rating the confidence of using the device correctly and confidence in the device delivering the correct full dose | At week 12
  Rating score on a 5-point Likert-type response scale. 1=Not at all confident, 5=Extremely confident.
Participant rating ease to learn how to use the device | At week 12
  Rating score on a 5-point Likert-type response scale. 1=Very difficult, 5=Very Easy.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (11):
- Poland (11):
  - Ginemedica Sp. z o.o. Sp.k, Wroclaw, Kuyavian-Pomeranian Voivodeship
  - CenterMed Krakow Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Diabetolog praktyka lekarska - Bartosz Bednarkiewicz, Lubin, Lower Silesian Voivodeship
  - Centrum Medyczne Ekamed sp. z o.o., Lublin, Lublin Voivodeship
  - Gabinet Lekarski Internistyczny Iwona Towpik, Zielona Góra, Lubusz Voivodeship
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji - Klinika Chorob Wewnetrznych, Endokrynologii i Diab, Warsaw, Masovian Voivodeship
  - Diabetica sp. z o.o., Nysa, Opole Voivodeship
  - Poradnia Diabetologiczna. Niepubliczny Zaklad Opieki Zdrowotnej Lege Artis, Bialystok, Podlaskie Voivodeship
  - NZOZ Gdanska Poradnia Cukrzycowa Sp. z o.o, Gdansk, Pomeranian Voivodeship
  - "Santa Familia PTG tódz, Lodz, Pomeranian Voivodeship
  - Diab Serwis POPENDA Spólka Jawna, Chorzów, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com